CLINICAL TRIAL: NCT06793566
Title: Effect of Tendon Vibrations on Motor Recovery of the Upper Limb in the Acute Phase of Stroke
Brief Title: Focal Muscle Vibrations in Acute Stroke
Acronym: VIBRAMAIN2
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Reorganisation and difficulties of neurology service of CHU Orleans
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHUO-2024-13
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Acute Stroke
Keywords: Acute stroke; Repetitive tendinous vibrations; Motor recovery; Non pharmacological therapy; Bedside intervention
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Each patient undergoes clinical evaluations at all time points by an experienced investigator blinded to group allocation and distinct from the recruiting personnel.
  Physical therapists, blinded to treatment allocation, are instructed on the duration, frequency, and content of therapy to ensure consistency across groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Vibration (Experimental): VG participants undergo rMV treatment, carried out for three consecutive days by 2 trained physiatrists; each daily session consists of three 10-minute treatment (impaired upper limb), interspersed with a 1-minute break. During the rMV, subjects are required to make a voluntary isometric contraction of the treated muscle
  Interventions: Device: Repeated Muscle Vibration (rMV)
- Control group (CG) (Sham Comparator): Participants in the CG undergo sham rMV, where the vibrator is positioned near the tendon but does not produce vibrations. Sham rMV treatment is carried out for three consecutive days by 2 trained physiatrists; each daily session consists of three 10-minute treatment (impaired upper limb), interspersed with a 1-minute break. During the rMV, subjects are required to make a voluntary isometric contraction of the treated muscle
  Interventions: Device: Repeated Muscle Vibration (rMV)

INTERVENTIONS:
Device: Repeated Muscle Vibration (rMV) — rMV treatment, carried out for three consecutive days by 2 trained physiatrists; each daily session consists of three 10-minute treatment (impaired upper limb), interspersed with a 1-minute break. During the rMV, subjects are required to make a voluntary isometric contraction of the treated muscle

SUMMARY:
A prospective, randomized, double-blind, sham-controlled trial designed to evaluate the effects of Repeated Muscle Vibration (rMV) on motor recovery in acute stroke patients treated within 72 hours of symptom onset

DETAILED DESCRIPTION:
After enrollment (T0), patients are randomly assigned to either the vibration group (VG) or the control group (CG). Patients in the VG will receive rMV treatment, while those in the CG receive sham treatment. Both interventions are administered on the 1st, 2nd, and 3rd days post-enrollment. Physiokinesitherapy (PT) and occupational therapy (OT) are provided daily to all patients, starting immediately after the T0 clinical evaluation. Patients are re-evaluated after 4 ± 1 days (T-1), marking the end of the treatment period.

Upon admission, demographic details and medical histories of all participants are recorded. Each patient undergoes clinical evaluations at all time points by an experienced investigator blinded to group allocation and distinct from the recruiting personnel. The clinical assessment includes stroke severity evaluation using the NIH Stroke Scale, motor and functional limb abilities using the Fugl-Meyer scale, SAFE score, and Motricity Index. Additionally, bioimpedance analysis of muscle mass and phase angle in the impaired upper limb is performed using the BWA device.

All participants follow a standardized daily rehabilitation program. Physical therapists, blinded to treatment allocation, are instructed on the duration, frequency, and content of therapy to ensure consistency across groups.

Low-amplitude rMV (frequency: 100 Hz; amplitude: 1-2 mm) is applied to the flexor carpi radialis and biceps brachii for upper limb treatment, using a commercial device (VibraMoov Physio, TechnoConcept, Mane, France). The rMV sessions are conducted over three consecutive days by two trained physiotherapists, with each daily session comprising three 10-minute treatments (per treated limb) interspersed with 1-minute breaks.

During the rMV sessions, participants are instructed to perform voluntary isometric contractions of the treated muscle. In contrast, CG participants undergo sham rMV, where the vibrator is positioned near the tendon but without vibration.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary patients in the acute phase of a sylvian ischemic stroke (from day 1 to day 7 post-stroke)
2. Estimated hospital stay expected to exceed 7 days
3. Age ≥ 18 years
4. Able to understand and follow evaluation instructions
5. Provided informed consent
6. Affiliated with a social security scheme
7. SAFE score between 4 and 7 on the affected side

Exclusion Criteria:

1. Individuals under guardianship or curatorship
2. Individuals deprived of liberty
3. Individuals under legal protection (safeguard of justice)
4. Other neurological or rheumatological conditions limiting mobility
5. Drowsiness (related to stroke or medication)
6. Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Upper limb Fugl Meyer Assessment Score (UL-FMA) | Day 4 from start of experiment
  This is a 66-point scale. A score of 0 corresponds to the maximum deficit and a score of 66 to a normal value.

SECONDARY OUTCOMES:
Upper limb strength | Day 4 from start of experiment
  A digital Jamar dynamometer is used to measure the flexion muscular strength of the deficient limb. The force value to be collected at each time point is the average of the 3 tests.Handgrip strength in kilograms
Motricity Index (Demeurisse) | Day 4 from start of experiment
  It assesses the motor skills of the upper limb as a whole, with elementary movements (thumb-index pinch,elbow flexion, shoulder abduction). Scoring ranges from 0 - corresponding to no movement - to 33 - corresponding to movement with normal strength. The upper limb score is calculated by summing the score obtained for each of the 3 movements, adding 1 and dividing by 100.
SAFE Score | Day 4 from start of experiment
  This is a 10 point scale. A score of 0 corresponds to no muscle contraction and a score of 10 to a normal muscular strength
Total NIHSS | Day 4 from start of experiment
  A 15-item impairment rating scale designed to assess the neurological consequences and degree of recovery of a stroke patient.
  Each item is rated from 0 to 2, 0 to 3 or 0 to 4. Each item that is non-testable is scored as "NT". A score of 0 indicates normal performance.
  NIHSS total scores range from 0 to 42, with higher values reflecting more severe brain damage.
muscular mass of the impaired upper limb | Day 4 from start of experiment
Phase angle of the impaired upper limb | Day 4 from start of experiment

CONTACTS AND LOCATIONS:
Overall Officials: Canan OZSANCAK, MD, Principal Investigator — CHU Orleans
Locations (1):
- CHU d'ORLEANS, Orléans, France

REFERENCES:
- [Background] Bertrand AM, Fournier K, Wick Brasey MG, Kaiser ML, Frischknecht R, Diserens K. Reliability of maximal grip strength measurements and grip strength recovery following a stroke. J Hand Ther. 2015 Oct-Dec;28(4):356-62; quiz 363. doi: 10.1016/j.jht.2015.04.004. Epub 2015 May 9. PMID 26206167
- [Background] Bobos P, Nazari G, Lu Z, MacDermid JC. Measurement Properties of the Hand Grip Strength Assessment: A Systematic Review With Meta-analysis. Arch Phys Med Rehabil. 2020 Mar;101(3):553-565. doi: 10.1016/j.apmr.2019.10.183. Epub 2019 Nov 13. PMID 31730754
- [Background] Caliandro P, Celletti C, Padua L, Minciotti I, Russo G, Granata G, La Torre G, Granieri E, Camerota F. Focal muscle vibration in the treatment of upper limb spasticity: a pilot randomized controlled trial in patients with chronic stroke. Arch Phys Med Rehabil. 2012 Sep;93(9):1656-61. doi: 10.1016/j.apmr.2012.04.002. Epub 2012 Apr 13. PMID 22507444
- [Background] Celletti C, Sinibaldi E, Pierelli F, Monari G, Camerota F. Focal Muscle Vibration and Progressive Modular Rebalancing with neurokinetic facilitations in post- stroke recovery of upper limb. Clin Ter. 2017 Jan-Feb;168(1):e33-e36. doi: 10.7417/CT.2017.1979. PMID 28240760
- [Background] Costantino C, Galuppo L, Romiti D. Short-term effect of local muscle vibration treatment versus sham therapy on upper limb in chronic post-stroke patients: a randomized controlled trial. Eur J Phys Rehabil Med. 2017 Feb;53(1):32-40. doi: 10.23736/S1973-9087.16.04211-8. Epub 2016 Sep 6. PMID 27598342
- [Background] Demeurisse G, Demol O, Robaye E. Motor evaluation in vascular hemiplegia. Eur Neurol. 1980;19(6):382-9. doi: 10.1159/000115178. PMID 7439211
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616
- [Background] Toscano M, Celletti C, Vigano A, Altarocca A, Giuliani G, Jannini TB, Mastria G, Ruggiero M, Maestrini I, Vicenzini E, Altieri M, Camerota F, Di Piero V. Short-Term Effects of Focal Muscle Vibration on Motor Recovery After Acute Stroke: A Pilot Randomized Sham-Controlled Study. Front Neurol. 2019 Feb 19;10:115. doi: 10.3389/fneur.2019.00115. eCollection 2019. PMID 30873102
- [Background] Abe T, Yoshimura Y, Imai R, Yoneoka Y, Tsubaki A, Sato Y. Impact of Phase Angle on Physical Function in Patients with Acute Stroke. J Stroke Cerebrovasc Dis. 2021 Sep;30(9):105941. doi: 10.1016/j.jstrokecerebrovasdis.2021.105941. Epub 2021 Jun 30. PMID 34217068
- [Background] Abe T, Yoshimua Y, Imai R, Sato Y. A Combined Assessment Method of Phase Angle and Skeletal Muscle Index to Better Predict Functional Recovery after Acute Stroke. J Nutr Health Aging. 2022;26(5):445-451. doi: 10.1007/s12603-022-1777-9. PMID 35587756